CLINICAL TRIAL: NCT06853717
Title: Implementation of Therapy Together With Early Childhood Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2022-258
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Unilateral Cerebral Palsy
Keywords: Constraint Induced Movement Therapy; Pediatric Constraint Induced Movement Therapy; Early Childhood Intervention; Therapy Together
MeSH Terms: interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: pre- and post- assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy Togther (Experimental): Therapy Together is a parent led intensive pediatric constraint induced movement therapy (P-CIMT) program for young children (3 months-2 years 11 months) with unilateral cerebral palsy (UCP). The research team developed the Therapy Together program due to the lack of clinical uptake in use of CIMT with children with UCP, even though there is consistent and robust evidence that demonstrates a positive treatment effect with the intervention. Therapy Together is based on the evidence and active ingredients of P-CIMT with a primary focus on clinical utility and translation of research to clinical practice
  Interventions: Behavioral: Therapy Together

INTERVENTIONS:
Behavioral: Therapy Together — CIMT consists of retraining the preferred hand by covering the hand with a soft mitt to promote the use of the assisting hand. With consistent practice, a toddler or infant builds the fine and gross motor skills of their assisting hand and bilateral coordination skills.
  Other Names: Constraint Induced Movement Therapy

SUMMARY:
The purpose of this project is to conduct a pilot hybrid type two implementation and efficacy study on Therapy Together with Early Childhood Intervention using an explanatory mixed methods approach to evaluate the efficacy and implementation of Therapy Together. Therapy Together is a parent led intensive pediatric constraint induced movement therapy (P-CIMT) program for young children (3 months-2 years 11 months) with unilateral cerebral palsy (UCP). The research team developed the Therapy Together program due to the lack of clinical uptake in use of CIMT with children with UCP, even though there is consistent and robust evidence that demonstrates a positive treatment effect with the intervention. Therapy Together is based on the evidence and active ingredients of P-CIMT with a primary focus on utility and translation of research to clinical practice.

DETAILED DESCRIPTION:
The long-term research goal is to implement Therapy Together, a caregiver-led pediatric constraint induced movement therapy program we developed for infants and toddlers with unilateral cerebral palsy, within regular health care models globally. The objective of this proposal is to conduct a pilot study to evaluate the efficacy and implementation of the Therapy Together program within the State of Texas Early Childhood Intervention program by conducting a mixed method, hybrid type two implementation and efficacy study guided by the RE-AIM Framework focusing on reach, effectiveness, adoption, and implementation. The central hypothesis is that Therapy Together can be successfully implemented within the early intervention model resulting in clinically significant improvements in hand function, occupational performance, and development. The rationale for this hypothesis is that Therapy Together is an adapted version of an evidence-based intervention specifically developed for implementation within standard of care practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants were children three months to two years and eleven months old who presented with asymmetric hand use with risk of developing cerebral palsy (CP) or have already been diagnosed with CP that present with unilateral upper limb impairment. Inclusion criteria were children who visually attended to objects, showed interest in them, and tried to reach for or grasp objects with their impaired upper extremity were included in the study.

Exclusion Criteria:

* Exclusion criteria were children with uncontrolled epilepsy, significant visual impairment, severe behavior problems or unable to complete assessment protocol were not included in the study.

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Mini-Assisting Hand Assessment (Mini-AHA) | pre-intervention and immediate post-intervention
  A semi-structured assessment for unilateral CP measuring effectiveness in bimanual hand
Canadian Occupational Performance Measure (COPM) | pre-intervention and immediate post-intervention
  A semi-structured interview that allows caregivers to evaluate and prioritize their child's current participation in the areas of self-care, leisure, and play
Developmental Assessment of Young Children, Second Edition (DAYC-2) | pre-intervention and immediate post-intervention
  The DAYC-2 is a normative-based assessment to identify children from birth to 5 years of age to assess a child's ability in areas of cognition, communication, social-emotional development, physical development, and adaptive behavior
Measure of Hand and Arm Performance | pre-intervention and immediate post-intervention
  The measure of hand and arm performance is an observation-based assessment of upper extremity movements developed by the researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Woman's Univeristy, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong RW. Definition and classification of cerebral palsy. Dev Med Child Neurol. 2007 Mar;49(3):166. doi: 10.1111/j.1469-8749.2007.00166.x. No abstract available. PMID 17355470
- [Background] Cioni G, D'Acunto G, Guzzetta A. Perinatal brain damage in children: neuroplasticity, early intervention, and molecular mechanisms of recovery. Prog Brain Res. 2011;189:139-54. doi: 10.1016/B978-0-444-53884-0.00022-1. PMID 21489387
- [Background] Creswell, J. W., & Creswell, J. D. (2018). Research design: Qualitative, quantitative, and mixed methods approaches. (5th ed). Sage Publications, 267-276.
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- [Background] Eliasson AC, Nordstrand L, Ek L, Lennartsson F, Sjostrand L, Tedroff K, Krumlinde-Sundholm L. The effectiveness of Baby-CIMT in infants younger than 12 months with clinical signs of unilateral-cerebral palsy; an explorative study with randomized design. Res Dev Disabil. 2018 Jan;72:191-201. doi: 10.1016/j.ridd.2017.11.006. Epub 2017 Nov 23. PMID 29175749
- [Background] Eliasson AC, Ullenhag A, Wahlstrom U, Krumlinde-Sundholm L. Mini-MACS: development of the Manual Ability Classification System for children younger than 4 years of age with signs of cerebral palsy. Dev Med Child Neurol. 2017 Jan;59(1):72-78. doi: 10.1111/dmcn.13162. Epub 2016 Jun 8. PMID 27273427
- [Background] Lidbeck C, Habel H, Martinsson C, Pettersson K, Lowing K. Motor Development in Children with Cerebral Palsy in Sweden-A Population-Based Longitudinal Register Study. Children (Basel). 2023 Nov 28;10(12):1864. doi: 10.3390/children10121864. PMID 38136066
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Palisano, R., Rosenbaum, P., Bartlett, D., & Livingston, M. (2007). Gross Motor Classification System expanded and revised. CanChild Centre for Childhood Disability Research. Retrieved on July 1, 2023 from https://canchild.ca/system/tenon/assets/attachments/000/000/058/original/GMFCS-ER_English.pdf
- [Background] Ramey SL, DeLuca SC, Stevenson RD, Conaway M, Darragh AR, Lo W; CHAMP. Constraint-Induced Movement Therapy for Cerebral Palsy: A Randomized Trial. Pediatrics. 2021 Nov;148(5):e2020033878. doi: 10.1542/peds.2020-033878. Epub 2021 Oct 14. PMID 34649982
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Sakzewski L, Ziviani J, Boyd RN. Efficacy of upper limb therapies for unilateral cerebral palsy: a meta-analysis. Pediatrics. 2014 Jan;133(1):e175-204. doi: 10.1542/peds.2013-0675. Epub 2013 Dec 23. PMID 24366991
- [Background] Saleh MN, Korner-Bitensky N, Snider L, Malouin F, Mazer B, Kennedy E, Roy MA. Actual vs. best practices for young children with cerebral palsy: a survey of paediatric occupational therapists and physical therapists in Quebec, Canada. Dev Neurorehabil. 2008 Jan-Mar;11(1):60-80. doi: 10.1080/17518420701544230. PMID 17943507
- [Background] Shierk, A., Roberts, H., Dubberly, K., Clegg, N. J., Fagan, M., Baldwin, D., Reyes, F., VanPelt, J., & Delgado, M. R. (2023). Therapy together: A caregiver led constraint induced movement therapy program for preschool aged children utilizing a virtual environment due to COVID 19. Journal of Occupational Therapy, Schools, and Early Intervention, 16(1), 39-50. https://doi.org/10.1080/19411243.2021.2003738
- [Background] Squires A, Sadarangani T, Jones S. Strategies for overcoming language barriers in research. J Adv Nurs. 2020 Feb;76(2):706-714. doi: 10.1111/jan.14007. Epub 2019 Jun 17. PMID 30950104
- [Background] Svensson K, Sundelin H, Eliasson AC. Outcomes of a Parent-Delivered Baby-mCIMT Model for Infants at High Risk of Unilateral Cerebral Palsy Using Remote Coaching in Telerehabilitation. Children (Basel). 2024 Jan 15;11(1):101. doi: 10.3390/children11010101. PMID 38255414
- [Background] Texas Health and Human Services Commission. (n.d.). Early childhood intervention services (ECI). Retrieved on July 1, 2023 from https://www.hhs.texas.gov/services/disability/early-childhood-intervention-services-eci
- [Background] U.S. Census Bureau. (2022). Limited English speaking households. American Community Survey, ACS 1-Year Estimates Subject Tables, Table S1602. https://data.census.gov/table/ACSST1Y2022.S1602?t=Language Spoken at Home&g=040XX00US48
- [Background] World Health Organization. (2007). International classification of functioning, disability and health, children & youth version (ICF-CY). World Health Organization. https://www.who.int/standards/classifications/international-classification-of-functioning-disability-and-health